CLINICAL TRIAL: NCT06829680
Title: Investigation of the Effects of Pilates Training Combined with Whole Body Vibration on Balance and Mobility in Individuals with Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Arzu Güçlü Gündüz, Profesor Doctor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-1602
Record Dates: First submitted 2025-02-08; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: Balance; Multiple Sclerosis; Mobility; Pilates; Vibration
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pilates-WBV (Experimental): 17 participants received Pilates and WBV training twice a week for 6 weeks. In each training session, the participants rested for 10 minutes between Pilates and WBV training.
  Interventions: Other: Pilates; Other: Whole Body Vibration
- Pilates (Active Comparator): 17 participants received Pilates training twice a week for 6 weeks
  Interventions: Other: Pilates

INTERVENTIONS:
Other: Pilates — The participants were given a total of 12 sessions of Pilates training, applied twice a week for 6 weeks, and each session lasted approximately 60 minutes. The 60-min session consisted of warm up and cool down (5 min each) and the main active phase (50 min).
  In the main active phase; "One leg stretch", "Double leg stretch", "One leg circle", "Heels together toes apart", "Shoulder bridge", "The hundreds", "Chest lift", "Criss cross", "Clam", "Side bend", "Arm opening", "Cobra", "Breast stroke", "Swimming", "Modified push-up", "Plank", "Leg pull prone" and "Squat" exercises were performed. The exercises were applied with 10 repetitions in the first 3 weeks and with 20 repetitions in the last 3 weeks.
Other: Whole Body Vibration — The participants were given a total of 12 sessions of WBV training, applied twice a week for 6 weeks.
  The vibration parameters were set as frequency: 20 Hz, amplitude: 2-3 mm, duration: 30-60 s and rest period: 60 s. The application time of the WBV training was 30 s for the first two weeks, 45 s for the next two weeks and 60 s for the last two weeks.
  The individuals were asked to maintain squat, shoulder bridge and quadruped positions statically for the first two weeks. Starting from the third week, they were asked to perform reciprocal upper extremity flexion and extension movements during the positions. The application was repeated 3 times in each position.
  Arms: Pilates-WBV

SUMMARY:
The aim of this study is to investigate the effects of Pilates training combined with whole-body vibration (WBV) on balance and mobility in individuals with Multiple Sclerosis (MS). The main questions it aims to answer are:

* Are the improvements in core stability, lower limb functional muscle strength, balance and mobility obtained with Pilates training combined with WBV (Pilates-WBV) in individuals with MS greater than with Pilates training alone?
* Are the improvements in upper extremity performance and fatigue obtained with Pilates-WBV training in individuals with MS greater than with Pilates training alone?

Researchers will compare Pilates-WBV training with a group that received Pilates training alone to see if there is any additional benefit.

Participants will:

* Take Pilates-WBV or Pilates training twice a week for 6 weeks
* Be evaluated with pre- and post-training

ELIGIBILITY:
Inclusion Criteria:

* Definitive Multiple Sclerosis diagnosed by a specialist
* Expanded Disability Status Scale (EDSS) score between 0-5
* Accepting participation in the study voluntarily

Exclusion Criteria:

* An MS attack within the last three months
* Pregnancy
* Endoprosthesis or electronic implant
* A cardiovascular, pulmonary or orthopedic disease
* A disease that can affect the immune system, such as infection or cancer
* Additional neurological disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
The Activities-specific Balance Confidence Scale | From enrollment to the end of treatment at 6 weeks
  The Activities-specific Balance Confidence Scale (ABC) evaluates balance confidence in daily living activities and includes 16 activities related to balance. Participants were asked to rate their perceived safety while performing these activities and their perceived risk of falling on a scale from 0 (completely unsafe) to 100 (completely safe). The total score is calculated by dividing the score by 16 and ranges from 0 to 100. Scores closer to zero indicate greater balance impairment and a higher risk of falls.
The Five Times Sit-to-Stand Test | From enrollment to the end of treatment at 6 weeks
  Lower extremity functional muscle strength was assessed by the Five Times Sit-to-Stand Test. The individuals were seated in a standard chair with arm support of 43-45 cm height, with their arms crossed on their chests. When the command "Start" was given, individuals were asked to stand up as quickly as possible and sit down and stand up 5 times. The score was the total time in seconds to complete the task. In the study, the test was repeated twice and the shortest time was recorded.
The Timed Up and Go Test | From enrollment to the end of treatment at 6 weeks
  Functional mobility was assessed by the Timed Up and Go Test (TUG). During the test, the individuals were asked to get up from the chair, walk 3 meters, turn around, walk back to the chair, and sit down. The score was the total time in seconds to complete the task. In the study, the test was repeated three times, and the average time was recorded.
The 6-Minute Walk Test | From enrollment to the end of treatment at 6 weeks
  Walking performance and functional exercise capacity were assessed using the Six-Minute Walk Test (6-MWT). Participants were instructed to walk at the highest speed they felt safe in a 30-meter straight pathway for six minutes. The score was the total walking distance in meters at the end of the test.
The Limits of Stability Test | From enrollment to the end of treatment at 6 weeks
  The Limits of Stability Test was assessed with The Biodex-Biosway Portable Balance System (Biodex Medical System Inc., Shirley, NY, USA). During the test, the individuals were asked to move their bodies toward target points displayed on the screen without lifting their feet and then return to the center point. During this movement, they were instructed to move as quickly and accurately as possible. The test results in a total percentage score. A lower score indicates decreased stability limits.
The Postural Stability Test | From enrollment to the end of treatment at 6 weeks
  The Postural Stability Test was assessed with The Biodex-Biosway Portable Balance System (Biodex Medical System Inc., Shirley, NY, USA). The test evaluates static balance by assessing the individual's ability to maintain their center of gravity over the support surface while standing. During the test, the individuals were asked to stand as still as possible. The test duration was 30 seconds and a total stability index score was calculated. The stability index scores range from 0 to 4, with lower scores indicating good postural stability.
The Modified Sensory Organization Test | From enrollment to the end of treatment at 6 weeks
  The Modified Sensory Organization Test (MSOT) was assessed with the Biodex-Biosway Portable Balance System (Biodex Medical System Inc., Shirley, NY, USA). In the test, by selectively disrupting visual and somatosensory inputs, it is determined which sensory inputs the individual relies on the most to maintain postural stability. The MSOT was performed under four conditions in the study: eyes open on a firm surface, eyes closed on a firm surface, eyes open on a soft surface, and eyes closed on a soft surface. The individuals were instructed to maintain their balance in all conditions. The test duration was 30 seconds for each condition. The sway index scores were calculated at the end of the test. The sway index scores range from 0 to 4, with lower sway index scores indicating decreased postural sway.
The Side-bridge Test | From enrollment to the end of treatment at 6 weeks
  The side-bridge test was used to assess core muscle endurance. The individuals were positioned in a straight line, lying on their left or right side with their legs fully extended. The individuals were asked to lift their body on forearms and toes, and maintain this position for as long as possible. When the individual was unable to maintain the position, the test was terminated. The score was the total time in seconds to complete the task. In the study, the test was performed twice, and the longer duration was recorded.
The Biering-Sorensen Test | From enrollment to the end of treatment at 6 weeks
  The Biering-Sorensen test was used to assess core muscle endurance. In this test, the individuals were asked to lie prone on a workout bench, aligning their anterior superior iliac spine with the edge of the bench, allowing the upper body to extend over the edge. An assisting partner secured the individuals' knees, hips, and pelvis. The individuals were instructed to fold their arms across their chest and to hold this position for as long as possible. When the individual was unable to maintain the position, the test was terminated. The score was the total time in seconds to complete the task. In the study, the test was performed twice, and the longer duration was recorded.
The Trunk Flexor Test | From enrollment to the end of treatment at 6 weeks
  The trunk flexor test was used to assess core muscle endurance. The individuals were positioned in a sit-up position with their back resting against a wedge angled at 60° from the floor. After the wedge was removed, they were asked to maintain this position for as long as possible. When the individual was unable to maintain the position, the test was terminated. The score was the total time in seconds to complete the task. In the study, the test was repeated twice, and the longer duration was recorded.
The Prone Bridge Test | From enrollment to the end of treatment at 6 weeks
  The prone bridge test was used to assess core muscle endurance. In this test, the individuals were asked to raise their bodies in a prone position, supporting themselves on their forearms and toes with their elbows flexed, maintaining this position for as long as possible. When the individual was unable to maintain the position, the test was terminated. The score was the total time in seconds to complete the task. In the study, the test was repeated twice, and the longer duration was recorded.
The Sit-ups Test | From enrollment to the end of treatment at 6 weeks
  The sit-ups test was used to assess core muscle strength. The test began when the individuals were instructed to ''go'', and they were asked to lift their upper body off the floor, raising the lower corner of the scapula. The score was recorded as the number of repetitions completed in 30 seconds. In the study, the test was performed twice, and the highest number of repetitions was recorded.
The Modified Push-ups Test | From enrollment to the end of treatment at 6 weeks
  The modified push-ups test was used to assess core muscle strength. The individuals were positioned on their hands and knees with hands shoulder-width apart and elbows fully extended. They dropped their hips and moved their hands forward until they created a straight line and a straight back from the knees to the hips to the shoulders. During the test, the individuals were asked to maintain this straight position while lowering their upper body until their elbows were bent to 90°, then pushing back up to the starting position. The score was recorded as the number of repetitions completed in 30 seconds. In the study, the test was performed twice, and the highest number of repetitions was recorded.

SECONDARY OUTCOMES:
The Nine-Hole Peg Test | From enrollment to the end of treatment at 6 weeks
  Upper extremity performance was assessed using the Nine-Hole Peg Test (9-HPT). The 9-HPT consists of a pegboard with 9 holes and 9 wooden pegs. Individuals were asked to place and remove all 9 pegs one at a time as fast as possible. The score was the total time in seconds to complete the task. In the study, the test was repeated twice for each extremity, and the average time was recorded for each side.
The Fatigue Severity Scale | From enrollment to the end of treatment at 6 weeks
  The Fatigue Severity Scale (FSS) assesses the severity of fatigue in the last month. It consists of 9 items, and the items are scored from 1 (strongly disagree) to 7 (strongly agree). The mean of the nine item scores is used as the FSS score. The scores that can be obtained from the test are between 1 and 7, and high scores indicate the presence of fatigue.
The Fatigue Impact Scale | From enrollment to the end of treatment at 6 weeks
  The Fatigue Impact Scale (FIS) assesses the impact of fatigue on physical, cognitive, and psychosocial functions in the last four weeks. It consists of 40 questions, with responses ranging from 0 (no problem) to 4 (extreme problem). The scores that can be obtained from the test are between 0 and 160, and high scores indicate a greater fatigue effect.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu GUCLU GUNDUZ, Professor Doctor, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Faculty of Health Science, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbasi M, Kordi Yoosefinejad A, Poursadeghfard M, Parsaei Jahromi F, Motealleh A, Sobhani S. Whole body vibration improves core muscle strength and endurance in ambulant individuals with multiple sclerosis: A randomized clinical trial. Mult Scler Relat Disord. 2019 Jul;32:88-93. doi: 10.1016/j.msard.2019.04.028. Epub 2019 Apr 30. PMID 31071658